CLINICAL TRIAL: NCT01292057
Title: Impulsivity and Drinking/Craving: Effect of a Dopamine Stabilizer Medication
Brief Title: Aripiprazole Effects on Alcohol Drinking and Craving
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Raymond F. Anton, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIH P50 AA010761; P50AA010761 (NIH)
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Alcohol Dependence
Keywords: Alcohol; Aripiprazole; Impulsivity; Alcoholism; drinking; treatment; craving; brain imaging; genetics
MeSH Terms: conditions — Alcoholism; Impulsive Behavior | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Active Comparator): Medication
  Interventions: Drug: Aripiprazole
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole(up to 15 mg/day) for 8 days
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Placebo — Placebo to match active drug Aripiprazole for 8 days
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether aripiprazole (marketed dopamine stabilizer) is effective in reducing of alcohol craving and drinking compared to placebo depending on participant's baseline level of impulsivity.

DETAILED DESCRIPTION:
Non-treatment seeking individuals meeting criteria for alcohol dependence (N=120) will be recruited through advertisement and paid for their participation. Subjects will have blood drawn for DNA analysis of various brain dopamine system genes. Alcoholics, after baseline evaluation, will be assigned through urn randomization to one of two experimental groups, depending on their baseline level of impulsivity, in which they will receive either aripiprazole (up to 15 mg/day) or an identical placebo. Subjects will take the study drug or placebo for 8 days (day 1-6 being the natural observation period). After a minimum of 24 hours of abstinence from alcohol (day 7-8) they will undergo an alcohol administration (priming dose) and motivated free choice drinking procedure (on day 8). Alcoholic subjects will receive a brief counseling session at the end of the study to enhance their awareness of problem drinking and to motivate them to seek treatment. Referral for treatment will be offered.

Each subject will undergo a functional MRI (functional magnetic resonance imaging) brain scan with cue stimulation on day 7, on the evening before the alcohol administration paradigm. fMRI (functional magnetic resonance) imaging brain imaging technology will be used to determine if alcoholics treated with aripiprazole differ in alcohol cue-induced activity in the nucleus accumbens. It is hypothesized that aripiprazole will reduce nucleus accumbens activation to alcohol cues compared to placebo.

Whether dopamine system genetic differences will be predict drinking, nucleus accumbens activity, and aripiprazole response will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 - 40 (to focus on an age group still on a trajectory of increasing alcohol consumption).
2. Meets the DSM IV criteria for current alcohol dependence including criterion 3 and/or 4 "loss of control over drinking" or "the inability to cut-down or stop drinking".
3. Currently not engaged in, and does not want treatment for, alcohol related problems.
4. Able to read and understand questionnaires and informed consent.
5. Lives within 50 miles of the study site.
6. Able to maintain abstinence for two days (without the aid of detoxification medications) as determined by self report and breathalyzer measurements.

Inclusion for fMRI (functional magnetic resonance imaging) Imaging:

1. Does not have metal objects in the head/neck.
2. Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

1. Currently meets DSM IV criteria for any other psychoactive substance dependence disorder.
2. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine THC (tetrahydrocannabinol) levels.
3. Meets DSM IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders and eating disorders, any other psychotic disorder or organic mental disorder.
4. Has current suicidal ideation or homicidal ideation.
5. Need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications and medications for ADHD (attention deficit hyperactivity disorder .
6. Currently taking medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, topiramate).
7. Clinically significant medical problems such as cardiovascular, renal, GI, or endocrine problems that would impair participation or limit medication ingestion.
8. Past history of alcohol related medical illness such as gastrointestinal bleeding, pancreatitis, peptic ulcer, hepatic cirrhosis or alcoholic hepatitis.
9. Hepatocellular disease indicated by elevations of SGPT (ALT) or SGOT (AST) greater than 2.5 times normal at screening.
10. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
11. Has current charges pending for a violent crime (not including DUI (Driving Under Intoxication) related offenses).
12. Does not have a stable living situation.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Anton, M.D., Principal Investigator — Medical University of South Carolian
Locations (1):
- Medical University of South Carolina, Institute of Psychiatry, Center for Drug and Alcohol Programs, Charleston, South Carolina, United States

REFERENCES:
- [Background] Anton RF, Schacht JP, Voronin KE, Randall PK. Aripiprazole Suppression of Drinking in a Clinical Laboratory Paradigm: Influence of Impulsivity and Self-Control. Alcohol Clin Exp Res. 2017 Jul;41(7):1370-1380. doi: 10.1111/acer.13417. Epub 2017 Jun 5. PMID 28493623
- See also: Alcoholism — http://www.nlm.nih.gov/medlineplus/
- See also: Ethanol — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: Aripiprazole — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: Clinical trials — http://clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole | Sugar Pill
Started | 49 | 50
Completed | 47 | 48
Not Completed | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Sugar Pill | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (5.6) | 27.0 (5.3) | 26.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 36 | 37 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Drinks Per Day During Natural (Usual Environment) Conditions
Description: "Natural" alcohol consumption period -- drinks per day consumed during the 6-day observation period
Time Frame: 6-day observation period
Measure: Mean (Standard Error); unit: standard drinks
Arm/Group | Aripiprazole | Sugar Pill
Number analyzed (Participants) | 47 | 48
standard drinks | 5.8 (0.4) | 6.4 (0.4)

2. Primary Outcome: Total Number of Drinks Consumed in Bar Lab
Description: This measure refers to a "bar lab" paradigm in which individuals received an initial "priming" drink of alcohol, targeted to produce a breath alcohol concentration (BrAC) of 30 mg%, and could then choose to consume up to 8 additional drinks, each targeted to produce a BrAC of 15 mg%, during the subsequent 2 hours. Thus, the total number of drinks consumed could range between 0 and 8.
Time Frame: 2 hours during the bar lab paradigm
Measure: Mean (Standard Error); unit: bar lab drinks
Arm/Group | Aripiprazole | Sugar Pill
Number analyzed (Participants) | 47 | 48
bar lab drinks | 3.3 (0.4) | 4.5 (0.4)

ADVERSE EVENTS:
Time Frame: 8 days
Description: Adverse event defined as any symptom rated "moderate" or "severe" on a 21-item physical symptom checklist. Items from the checklist were: trouble sleeping, daytime sleepiness, nervousness, irritability, trouble concentrating, feeling depressed, abdominal pain, nausea/vomiting, constipation, joint pain, headache, dizziness, low energy, skin rash, ears ringing, vision blurry, itching, increased libido, decreased libido, difficulty reaching orgasm, and inability to reach orgasm.
Arm/Group | Aripiprazole | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 39/47 | 17/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=47) | Sugar Pill (N=48)
Trouble sleeping (Nervous system disorders) | 14 | 9
Daytime sleepiness (Nervous system disorders) | 31 | 8
Nervousness (Nervous system disorders) | 4 | 1
Irritability (Nervous system disorders) | 8 | 6
Trouble concentrating (Nervous system disorders) | 14 | 3
Feeling depressed (Psychiatric disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 0
Low energy (Nervous system disorders) | 22 | 0
Increased libido (Reproductive system and breast disorders) | 3 | 2
Decreased libido (Reproductive system and breast disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No